CLINICAL TRIAL: NCT07062887
Title: A Digital Mindfulness and Biometric Feedback Application for Young Adults With Type 1 Diabetes
Brief Title: Digital Mindfulness for Young Adults With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000039191
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes (T1D); Diabetes Secondary to Pancreatitis
Keywords: mindfulness; stress; sleep; smartwatch; sensors
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness App (Experimental): Use the mindfulness app for 6 weeks, wear an actigraphy watch, share the data from your own continuous glucose monitor (CGM), answer surveys and interviews about the app.
  Interventions: Behavioral: Mindfulness app

INTERVENTIONS:
Behavioral: Mindfulness app — Mindfulness app called Calm Health. It has mindfulness guidance modules related to different aspects of physical and mental health, including type 1 diabetes. It also provides a final report to help you track the relationship between mindfulness and your blood sugar, stress, and sleep.

SUMMARY:
The purpose of this research study is to test a mindfulness app called Calm Health among young adults with type 1 diabetes or other absolute insulin deficiency diabetes. Mindfulness is the practice of being aware of your thoughts and feelings in the moment without judgment or negative reaction. All participants will receive mindfulness guidance and personalized feedback about the relationship among your mindfulness, blood sugar, stress, and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving diabetes care at Yale New Haven Children's Hospital or Yale New Haven Hospital.
2. Sign and date informed consent form we will provide
3. Willingness to complete procedures and availability for duration of the study
4. Aged 18-30 years
5. Diagnosed with type 1 diabetes (T1D) or other absolute insulin deficiency diabetes (latent autoimmune diabetes of adulthood, diabetes secondary to pancreatitis) for at least 1 year.
6. User of a continuous glucose monitor (CGM) in your routine clinical care for at least the past 2 weeks.
7. Able to use a smartphone.
8. Able to read and write English.

Exclusion Criteria:

1. Current meditation or mindfulness practice meeting or exceeding the study's recommended schedule
2. Current severe untreated psychiatric illness (e.g., bipolar disorder, schizophrenia, major depression, panic disorder, borderline personality disorder, organic mood or mental disorders) or active suicidal ideation
3. New or unstable psychopharmaceutical treatment in past 2 months.
4. Current or planned pregnancy during study period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mindfulness app usage | 6 weeks
  Minutes of usage per week

SECONDARY OUTCOMES:
Exit survey | 6 weeks
  Likert-style survey of usability, acceptability, appropriateness, and feasibility. Responses are on a scale from 1 (very dissatisfied) to 5 (very satisfied)
T1D-related emotional distress | 6 weeks
  Problem Areas in Diabetes (PAID) scale. Responses are on a scale from 0 (Not a problem) to 4 (serious problem)
Type 1 Diabetes Distress | 6 weeks
  Type 1 Diabetes Distress Scale (T1-DDS). Consists of common distressing things about living with type 1 diabetes. Scores range from 1 (not a problem) to 6 (very serious problem).
Type 1 diabetes-specific health related quality of life | 6 weeks
  Type 1 diabetes and life (T1DAL) scale. Aspects of life with type 1 diabetes. Scores range from 1 (no, not true at all) to 5 (yes, very true).
Anxiety | 6 weeks
  Generalized anxiety disorder 7-question screener (GAD-7). Participants rate frequency of symptoms. Scores range from 0 (not at all) to 3 (nearly every day).
Depression | 6 weeks
  Patient Health Questionnaire 9-question screener. Participants rate frequency of symptoms. Scores range from 0 (not at all) to 3 (nearly every day).
Mindful attention awareness | 6 weeks
  Mindful attention awareness scale. Participants rate frequency of typical experiences. Scores range from 1 (almost always) to 6 (almost never).
Self-Compassion | 6 weeks
  Self-Compassion Scale. Participants rate frequency of behaviors. Scores range from 1 (almost always) to 5 (almost never).
Practice of mindfulness | 6 weeks
  Five-facet mindfulness questionnaire. Participants rate frequency of behaviors. Scores range from 1 (never or very rarely true) to 5 (very often or always true).

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Nally, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Survey scores, glucose, physical activity, sleep, heart rate, heart rate variability, respiratory rate
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Start date: Publication of primary manuscript End date: Indefinitely
Access Criteria: The data will be available immediately following publication, with no end dates. The data will be shared with researchers who provide a methodologically sound proposal to achieve the aims of the approved proposal. The proposals should be directed to Dr. Garrett Ash at Yale University (garrett.ash@yale.edu). To gain access, data requesters must sign a data access agreement.